CLINICAL TRIAL: NCT01033526
Title: A Two-arm, Multicenter, Randomized, Double-blind, Single Dose Placebo-controlled Parallel Groups Study Evaluating Efficacy and Tolerability of 800 mg Acetylsalicylic Acid (Aspirina® C) in Adult Patients With a Common Cold During a Two Hour in Patient Phase; and a Follow-up Period of Five Days of Home Treatment as Required
Brief Title: Symptomatic Treatment of Common Cold Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Consumer Care Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11756; EudraCT: 2004-004683-71
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-12

CONDITIONS: Common Cold
Keywords: Symptomatic treatment of Common Cold symptoms
MeSH Terms: conditions — Common Cold | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 1 (Experimental)
  Interventions: Drug: Aspirin (Acetylsalicylic acid, BAYE4465)

INTERVENTIONS:
Drug: Aspirin (Acetylsalicylic acid, BAYE4465) — 1-2 tablets Acetylsalicylic Acid 400 mg (in combination with Ascorbic Acid 240 mg) as needed every 4-6 hours over a maximum of 5 days
  Arms: Arm 1
Drug: Placebo — 1-2 tablets matching Placebo as needed every 4-6 hours over a maximum of 5 days
  Arms: Arm 2

SUMMARY:
A two-arm, multicenter, randomized, double-blind, single dose placebo-controlled parallel groups study evaluating efficacy and tolerability of 800 mg Acetylsalicylic Acid (Aspirina C) in adult patients with a common cold during a two hour in patient phase; and a follow-up period of five days of home treatment as required.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Onset of cold symptoms within 48 hours before screening
* Objective symptoms of common cold
* Subjective symptoms of common cold

Exclusion Criteria:

* Pregnancy or lactation period
* Active peptic ulcer
* Hemorrhagic diathesis
* History of chronic or recurrent ulcer disease or history of gastro-intestinal bleeding
* Hypersensitivity to acetylsalicylic acid, to paracetamol, to any other component of the study medication, to anti-inflammatory or antirheumatic drugs, to other allergens

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2005-10; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change in Cold Symptoms (patient Wisconsin Upper Respiratory Symptom Survey (WURSS domain 2 score) from baseline | 2 hours following intake of the first study medication dose

SECONDARY OUTCOMES:
Changes in Common Cold Profile (sum of WURSS domains 1 182 3) | At each of five evenings during the follow-up period (or directly prior to the first intake of rescue medication during the follow-up period)
Changes in Global Cold Severity (WURSS domain 1) | At each of five evenings during the follow-up period (or directly prior to the first intake of rescue medication during the follow-up period)
Changes in Cold Symptoms (WURSS domain 2) | At each of five evenings during the follow-up period (or directly prior to the first intake of rescue medication during the follow-up period)
Changes in Cold-specific Functional Impairments (WURSS domain 3) | At each of five evenings during the follow-up period (or directly prior to the first intake of rescue medication during the follow-up period)
Changes in Global Cold Severity (WURSS domain 4) | At each of five evenings during the follow-up period (or directly prior to the first intake of rescue medication during the follow-up period)
Adverse Event Collection | Until end of study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (28):
- Italy (28):
  - Borgo di Terzo, Bergamo
  - Brembate, Bergamo
  - Calusco d'Adda, Bergamo
  - Capriate San Gervasio, Bergamo
  - Caravaggio, Bergamo
  - Casazza, Bergamo
  - Cologno al Serio, Bergamo
  - Covo, Bergamo
  - Dalmine, Bergamo
  - Mozzanica, Bergamo
  - Ponte San Pietro, Bergamo
  - Seriate, Bergamo
  - Verdello, Bergamo
  - Vertova, Bergamo
  - Villa d'Adda, Bergamo
  - Angera, Varese
  - Carnago, Varese
  - Cavaria, Varese
  - Comerio, Varese
  - Cunardo, Varese
  - Fagnano Olona, Varese
  - Induno Olona, Varese
  - Sesto Calende, Varese
  - Solbiate Olona, Varese
  - Varese, Varese
  - Vedano Olona, Varese
  - Vergiate, Varese
  - Albano Sant'Alessandro